CLINICAL TRIAL: NCT02661360
Title: Effects of Swaddling During Bottle Feeding on Infants Born Preterm
Brief Title: Effects of Swaddling on Infants During Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-00493
Record Dates: First submitted 2016-01-20; First posted 2016-01-22 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Premature Birth
Keywords: swaddling
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Starting condition of swaddled (Experimental)
  Interventions: Behavioral: Swaddling Intervention for Preterm Infants; Behavioral: Unswaddled Control
- Starting Condition of Unswaddled (Experimental)
  Interventions: Behavioral: Swaddling Intervention for Preterm Infants; Behavioral: Unswaddled Control

INTERVENTIONS:
Behavioral: Swaddling Intervention for Preterm Infants — Procedure for swaddling includes folding one corner of the blanket down two thirds of the way down the blanket in order to make the blanket into a triangular shape. The infant will be positioned with shoulders at the fold of the blanket. The infant will be positioned with the blanket so that elbows, hips, and knees flexed with hands near the face by wrapping one side of the blanket across the chest holding the hands in place, pulling the bottom corner up toward the infant's face, and securing the blanket with the last corner pulled across the infant's chest again and around their back. The blanket will be tight enough to keep extremities in place but one finger will be able to be placed between the infant and the blanket.
Behavioral: Unswaddled Control — Procedure for control is blanket loosely draped across the infant without providing containment and without touching the anterior surface of the infant.

SUMMARY:
The purpose of this randomized, within-subject, cross-over study is to examine if swaddling affects bottle feeding performance in infants born preterm. Results from research will have implication on neurobehavioral and physiologic outcomes as important indicators for the possible effect of swaddling during bottle feeding.

DETAILED DESCRIPTION:
Once an infant is orally feeding a minimum of two times per nursing shift for four consecutive nursing shifts, the infant will be randomly assigned to receive the intervention (swaddling) or control condition (no swaddling) first, by the research OT randomly choosing an envelope with the assignment enclosed. The intervention and control feedings for each infant will be consecutive and will take place at the infant's bedside in the NICU. Infants will be assessed at each nursing care time for feeding readiness by the research OT and feeding OT according the policies of the NYU Langone Medical Center NICU, which utilizes the Infant-Driven Feeding Scale-Readiness (Appendix B) (Ludwig & Waitzman, 2006). When the infant demonstrates readiness, the first condition will be initiated. At the next feeding when the infant demonstrates readiness, the opposite condition will be applied. If the infant is not available due to procedures or not demonstrating feeding readiness, at the next two caregiving times after the first feeding, the infant will be discontinued for that day and will start the study over the next day.

ELIGIBILITY:
Inclusion Criteria:

* all infants born before 34 weeks gestational age will be included as long as they do not have any exclusion criteria
* infants born before 34 weeks gestational age is 33 weeks 3 days to 35 weeks 0 days, with attainment of exclusive bottle feeding at 36 weeks gestational age at the earliest.
* Infants who are multiples will be included but restricted to twins and triplets.
* Infants will only be included if their parents provide informed consent for participation of their infant in the study.

Exclusion Criteria:

The exclusion criteria are factors commonly associated with feeding problems in infants beyond prematurity, including:

* Infants who are exclusively breastfed
* Higher order multiples than twins and triplets (ie. quadruplets)
* Infants with conditions that may affect feeding performance:

  1. Grades III and IV intraventricular hemorrhage
  2. Necrotizing enterocolitis
  3. Congenital cardiac anomalies (except medically managed patent ductus arteriosus)
  4. Genetic syndromes
  5. Craniofacial abnormalities

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Oral feeding readiness measured by subtest of Early Feeding Skills Assessment (EFS) | 1 Day
Feeding engagement measured by subtest of Early Feeding Skills Assessment (EFS) | 1 Day
Oral motor organization measured by subtest of Early Feeding Skills Assessment (EFS) | 1 Day
Swallow coordination measured by subtest of Early Feeding Skills Assessment (EFS) | 1 Day
Physiologic stability measured by subtest of Early Feeding Skills Assessment (EFS) | 1 Day
  Stability of heart rate and respiratory rate are indicative of the ability of the infant born preterm to cope with stress during bottle feeding
Feeding recovery measured by subtest of Early Feeding Skills Assessment (EFS) | 1 Day
Number of significant changes in heart rate (bradycardia | 1 Day
Number of significant oxygen desaturations | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Steve Vanlew, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States